CLINICAL TRIAL: NCT04225975
Title: Evaluation of Cerebral, Hemodynamic and Neuronal Activities in Neonates in the Immediate Postpartum
Brief Title: Neonate Cerebral Activity in Immediate Post Partum
Acronym: POSTPARTUM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PI2019_843_0031
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Anoxia-Ischemia, Brain; Neonatal Encephalopathy
Keywords: Anoxia-Ischemia, Brain; postpartum; Electroencephalography; Cerebral oxymetry; Near Infrared spectroscopy; EEG; NIRS; Neonate
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Electroencephalography; Oximetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: electroencephalogram — Within the 5 min after birth the electroencephalogram of the neonates will be recorded with the aid of a patch on the scalp
Diagnostic Test: oxymetry — Within the 5 min after birth the cerebral oxymetry of the neonates will be recorded with the aid of a patch on the scalp

SUMMARY:
Neonatal anoxia-ischemia causes significant neurodevelopmental disorders. In this study the investigators want to better understand the interactions between the nervous and the hemodynamic cerebral systems during the adaptation of the neonate to ectopic life just after birth. Birth is an at risk situation of neonatal anoxic ischemia and the lack of objective criteria for cerebral tissue oxygenation has consequences on neuronal activity. Ph cord analysis is inadequate and only indirectly reflects the state of cerebral oxygenation. Both neuronal and vascular systems are part of the same functional entity and the analysis of their interactions is likely to reveal some early malfunctions of these networks.

In this study, the investigators want to develop a multi-scale, multimodal approach that allows simultaneous interrogation of both neuronal and vascular compartments during the 15 minutes after delivery. The investigators will record, with the aid of a single sensor placed on the scalp of the child, the electroencephalogram and the cerebral tissue oxygenation. The investigators will measure interactions by means of correlation analysis between both signals.

ELIGIBILITY:
Inclusion Criteria:

* Full term neonates between 36 and 41 weeks Gestational Age

Exclusion Criteria:

* Premature neonates
* Neonates of twin pregnancy
* Suspicion of congenital malformation seen in antenatal ultrasound
* Any pathology requiring pediatric care from birth
* Newborns whose mothers had a chronic viral infection such as AIDS, hepatitis B or C, or who had a multidrug-resistant bacteria

Ages: 1 Minute to 15 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Temporal correlation with EEG | within the 5 minutes after birth
  Within the 5 min after birth the electroencephalogram and the cerebral oxymetry of the neonates will be recorded with the aid of a patch on the scalp. A multimodal approach must be developed to interrogate the dynamics and interactions of neuronal and vascular compartments, which constitute a single functional unit.
time-frequency correlation with EEG | within the 5 minutes after birth
  Within the 5 min after birth the electroencephalogram and the cerebral oxymetry of the neonates will be recorded with the aid of a patch on the scalp. A multimodal approach must be developed to interrogate the dynamics and interactions of neuronal and vascular compartments, which constitute a single functional unit.
temporal correlation with NIRS signals | within the 5 minutes after birth
  Within the 5 min after birth the electroencephalogram and the cerebral oxymetry of the neonates will be recorded with the aid of a patch on the scalp. A multimodal approach must be developed to interrogate the dynamics and interactions of neuronal and vascular compartments, which constitute a single functional unit.
time-frequency correlation with NIRS signals | within the 5 minutes after birth
  Within the 5 min after birth the electroencephalogram and the cerebral oxymetry of the neonates will be recorded with the aid of a patch on the scalp. A multimodal approach must be developed to interrogate the dynamics and interactions of neuronal and vascular compartments, which constitute a single functional unit.

SECONDARY OUTCOMES:
Mode of delivery correlation with temporal and EEG data | within the 5 minutes after birth
  Within the 5 min after birth the electroencephalogram and the cerebral oxymetry of the neonates will be recorded with the aid of a patch on the scalp.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No